CLINICAL TRIAL: NCT04767542
Title: Bakirkoy Dr. Sadi Konuk Training and Research Hospital
Brief Title: Postoperative Pain Difference for 'IV Paracetamol' and TAP Block' in Acute Cholecystitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Turgut Donmez, Ass. Prof. Dr., Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Bakirkoy Sadi Konuk
Record Dates: First submitted 2021-02-05; First posted 2021-02-23 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Transversus Abdominis Plane (TAP) Block
Keywords: acute cholecystitis; postoperative pain; transversus abdominis plane block
MeSH Terms: conditions — Bites and Stings; Cholecystitis, Acute; Pain, Postoperative | interventions — Infusions, Intravenous; Acetaminophen; Anesthesia, Local

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paracetamol (Sham Comparator): Patients with emergency LC will be administered intravenously 1 gr vial of paracetemol in 30 minutes during the awakening phase.
  Interventions: Drug: Intravenous Infusion
- Transversus Abdominis Plane Block (Active Comparator): With USG, the lateral part of the latissumus dorsi muscle attaches to the external lip of the iliac crest, just behind the middle axillary line and the end is directed slightly cranially, first through the external oblique muscle and fascia, then the internal oblique muscle and fascia, and after hydrodissection with saline for about 15-20 ml of local anesthetic agent (Bupivacaine 0.5%) will be injected bilaterally
  Interventions: Procedure: Local anesthesia

INTERVENTIONS:
Drug: Intravenous Infusion — analgesic
  Other Names: Paracetamol
  Arms: Paracetamol
Procedure: Local anesthesia — Local anesthetic agent (Bupivacaine 0.5%) will be injected bilaterally to transverses abdominis muscle
  Arms: Transversus Abdominis Plane Block

SUMMARY:
Patients with acute cholecystitis or pancreatitis due to gallstones benefit from emergency laparoscopic cholecystectomy (LC). Patients with emergency LC show improvement in their quality of life within one month compared to those treated. Delayed LC (after the acute phase has passed and recovered) and less time to work. This strategy reduces the risk of repeated admissions with more pain or pancreatitis. There are many studies on the effectiveness of the Elective LC and Transversus Abdominis Plan (TAP) Block on pain. However, a prospective study on the reduction of postoperative pain with emergency LC and TAP Block has not been carried out until now. This study will be conducted to evaluate the effectiveness of the TAP Block in patients undergoing emergency LC.

DETAILED DESCRIPTION:
Patients to be included in the study will be selected from the group between the ages of 18 and 70 who apply to general surgery and emergency outpatient clinics, depending on patient approval. All patients will be informed about the surgery and procedures to be performed. Patients who agree to participate in the study will be included in the study. The study will be carried out by 2 surgeons with 5 years of laparoscopic cholecystectomy (LC) experience. Adult patients presenting with acute cholecystitis who underwent emergency LC by one of the two surgeons will be included in the study. These two surgeons will be responsible for participant registration. Patients with fever greater than 3.37.2 ℃, including 1) a diagnosis of acute cholecystitis confirmed by hepatobiliary ultrasound, 2) a high leukocyte count (> 7 × 109 / L), will be included in the study. Patients undergoing elective laparoscopic cholecystectomy (E-LC) and patients who are converted to an open procedure will be excluded from the study. Patients will be divided into two groups. In Group A, patients with emergency LC will be administered intravenously 1 gr vial of paracetemol in 30 minutes during the awakening phase. In Group B, the lateral part of the latissumus dorsi muscle attaches to the external lip of the iliac crest, behind the middle axillary line and the end is directed towards the cranial, firstly the external oblique muscle and fascia, then the internal oblique muscle and fascia, and after hydrodissection with saline physiological. 15-20 ml of local anesthetic agent (Bupivacaine 0.5%) will be injected bilaterally.

Standard laparoscopic cholecystectomy will be applied in two groups. Nasogastric tube will be inserted after intubation in both groups and will be removed at the end of the operation. Age, height, weight, ASA score, body mass index, duration of surgery, complications, comorbidities, fever, leukocyte, CRP levels, ALT, AST, GGT, total bilirubin, direct bilirubin values will be recorded. Pulse, heart rate, systolic and diastolic pressures, Oxygen saturation (with a palimeter) will be recorded during surgery in both groups. VAS and VRS pain scoring will be done after surgery. VAS (Visuale analogue score) 0-10 cm and VRS (no pain in cough (score = 0); pain in cough, not in deep breathing (score = 1); pain in deep breathing, but not at rest (score = 2); at rest pain will be evaluated as mild (score = 3); pain at rest, severe (score = 4)). Evaluations will be made statistically between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Acute stony cholecystitis
* Acute acalculous cholecystitis
* 18-70 years old

Exclusion Criteria:

* Open cholecystectomy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-03-15 (Estimated); Primary Completion 2021-09-15 (Estimated); Study Completion 2021-10-15 (Estimated)

PRIMARY OUTCOMES:
Pain Score | Preoperative 1th hour
  Postoperative Verbal Rating Score and Visuale analogue scoring will be done.

SECONDARY OUTCOMES:
Pain Score | Postoperative 1st hour
  Postoperative Verbal Rating Score will be done
Pain Score | Postoperative 4th hour
  Postoperative Verbal Rating Score and Visuale analogue scoring will be done.
Pain Score | Postoperative 8th hour
  Postoperative Verbal Rating Score and Visuale analogue scoring will be done.
Pain Score | Postoperative 12th hour
  Postoperative Verbal Rating Score and Visuale analogue scoring will be done.
Pain Score | Postoperative 24th hour
  Postoperative Verbal Rating Score and Visuale analogue scoring will be done.

CONTACTS AND LOCATIONS:
Overall Officials: Turgut Donmez, Ass. Prof., Study Director — Bakirkoy Sadi Konuk

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yahya Gumusoglu A, Ferahman S, Gunes ME, Surek A, Yilmaz S, Aydin H, Gezmis AC, Aliyeva Z, Donmez T. High-Volume, Low-Concentration Intraperitoneal Bupivacaine Study in Emergency Laparoscopic Cholecystectomy: A Double-Blinded, Prospective Randomized Clinical Trial. Surg Innov. 2020 Oct;27(5):445-454. doi: 10.1177/1553350620914198. Epub 2020 Apr 3. PMID 32242764
- [Result] Peng K, Ji FH, Liu HY, Wu SR. Ultrasound-Guided Transversus Abdominis Plane Block for Analgesia in Laparoscopic Cholecystectomy: A Systematic Review and Meta-Analysis. Med Princ Pract. 2016;25(3):237-46. doi: 10.1159/000444688. Epub 2016 Feb 16. PMID 26885872